CLINICAL TRIAL: NCT06364280
Title: Pediatric Prehospital Airway Resuscitation Trial
Acronym: Pedi-PART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Utah (Other)
Responsible Party: Principal Investigator, Henry Wang, MD, Professor, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023X0135; UG3HL165019 (NIH); U24HL165014 (NIH); UH3HL165019 (NIH); R01HL181356 (NIH)
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Heart Arrest, Out-Of-Hospital; Wounds and Injuries; Respiratory Insufficiency in Children; Child, Only; Critical Illness
Keywords: airway management; intubation, intratracheal; emergency medical services; children; heart arrest; injuries; respiratory insufficiency
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Wounds and Injuries; Critical Illness; Heart Arrest; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: The trial uses a Bayesian Adaptive Sequential Platform Trial (BASIC-PT) framework.
  The study interventions are strategies of prehospital airway management: [BVM-only], [BVM followed by SGA] and [BVM followed by ETI].
  The trial will be organized and executed in two successive stages. In Stage I of the trial, EMS personnel will alternate between two strategies: [BVM-only] or [BVM followed by SGA]. The [winner of Stage I] will advance to Stage II based upon results of Bayesian interim analyses. In Stage II of the trial, EMS personnel will alternate between [BVM followed by ETI] vs. [Winner of Stage I].
  The interventions will be quasi-randomized using alternate day assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- BVM-only (Active Comparator): Initial strategy of airway management using Bag-Valve-Mask (BVM) only.
  Interventions: Device: BVM
- BVM followed by SGA [BVM+SGA] (Active Comparator): Initial strategy of airway management using Bag-Valve-Mask (BVM) followed by Supraglottic Airway (SGA).
  Interventions: Device: BVM; Device: SGA
- BVM followed by ETI [BVM+ETI] (Active Comparator): Initial strategy of airway management using Bag-Valve-Mask (BVM) followed by Endotracheal Intubation (ETI).
  Interventions: Device: BVM; Device: ETI

INTERVENTIONS:
Device: BVM — Bag-Valve-Mask Ventilation
Device: SGA — Supraglottic Airway
  Arms: BVM followed by SGA [BVM+SGA]
Device: ETI — Endotracheal Intubation
  Arms: BVM followed by ETI [BVM+ETI]

SUMMARY:
This study is a Phase 3, multi-center, Bayesian Adaptive Sequential Platform Trial testing the effectiveness of different prehospital airway management strategies in the care of critically ill children. Emergency Medical Services (EMS) agencies affiliated with the Pediatric Emergency Care Applied Research Network (PECARN) will participate in the trial. The study interventions are strategies of prehospital airway management: [BVM-only], [BVM followed by SGA] and [BVM followed by ETI]. The primary outcome is 30-day ICU-free survival. The trial will be organized and executed in two successive stages. In Stage I of the trial, EMS personnel will alternate between two strategies: [BVM-only] or [BVM followed by SGA]. The [winner of Stage I] will advance to Stage II based upon results of Bayesian interim analyses. In Stage II of the trial, EMS personnel will alternate between [BVM followed by ETI] vs. [Winner of Stage I].

DETAILED DESCRIPTION:
Cardiac arrest, respiratory failure, and major trauma are devastating critical conditions in children. Resuscitation from critical illness requires skillful airway management to optimize the delivery of oxygen to the lungs, preventing irreparable damage to the brain and heart. As the first to provide resuscitation care for critically ill children, prehospital EMS personnel are often the first to perform life-saving airway management.

The most common prehospital airway management techniques (bag-valve-mask ventilation [BVM], endotracheal intubation [ETI], and supraglottic airway insertion [SGA]) have important trade-offs between risks and benefits. Despite the challenges of ETI and national recommendations favoring BVM, many EMS personnel favor ETI over BVM. Newer SGA devices such as the laryngeal tube (LT), laryngeal mask airway (LMA), and i-gel® have not been compared with other techniques in children. National organizations, including the Agency for Healthcare Research and Quality, have declared the need for new, rigorous trials of all techniques to determine the best strategies for prehospital airway management in children. Interviews with front-line EMS personnel underscore the dire need for clear and strategic guidelines for managing the pediatric airway.

The Pediatric Prehospital Airway Resuscitation Trial (Pedi-PART) will determine the best strategies for prehospital airway management in critically ill children. The trial aims are Aim I-Primary Objective (Effectiveness)-Stage I: Determine if [BVM-only] or [BVM followed by SGA] results in better ICU-free survival in critically ill children with cardiac arrest, major trauma, or respiratory failure. Stage II: Determine if [winner of Stage I] or [BVM followed by ETI] results in better ICU-free survival. Bayesian analyses will determine the transition from Stage I to Stage II, ensuring optimal deployment of available subjects to address the postulated questions. Aim 2- Secondary Objective (Safety)-Stage I: Determine if [BVM followed by SGA] results in fewer prehospital and hospital safety events compared with [BVM-only] in critically ill children with cardiac arrest, major trauma, or respiratory failure. Stage II: Determine if the winner of Stage I results in fewer safety events compared with [BVM followed by ETI].

The trial will use a Bayesian Adaptive Sequential Comparison Platform Trial (BASiC-PT) design and will be executed in two sequential stages. Stage I: Determine if [BVM-only] or [BVM followed by SGA] results in better ICU-free survival in critically ill children with cardiac arrest, major trauma, or respiratory failure. Stage II: Determine if [winner of Stage I] or [BVM followed by ETI] results in better ICU-free survival. Bayesian analyses will determine the transition from Stage I to Stage II, ensuring optimal deployment of available subjects to address the postulated questions.

ELIGIBILITY:
Inclusion criteria are:

* At least 24 hours old and <18 years old
* Cardiopulmonary arrest, major trauma or respiratory failure
* Life-saving care initiated or continued by Pedi-PART EMS personnel as part of an emergency "9-1-1" response
* Requiring active airway management (BVM or higher level of respiratory support

Exclusion criteria are:

* Prisoners
* Pre-existing tracheostomy
* Pre-existing do-not-resuscitate/do-not-intubate status
* Visibly or known to be pregnant
* Initial advanced airway attempt by an EMS agency not affiliated with the study
* Interfacility transports

EMS personnel will use bystander reports or follow local protocols to establish patient age and pregnancy status.

Ages: 24 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
30-day ICU-free survival | 30 days
  The number of days in the first 30 days after the treatment event where: 1) the patient was not known to have died; and 2) the patient was not hospitalized in the intensive care unit. ICU admission/discharge criteria will not be standardized.

SECONDARY OUTCOMES:
Neurologic outcome upon hospital discharge | Identified through end of study but no later than 30 days after final enrollment.
  Outcome will be measured with Pediatric Cerebral Performance Category score (PCPC - 1 = normal, 2 = mild disability, 3 = moderate disability, 4 = severe disability, 5 = coma or vegetative state, 6 = dead).

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Wang, MD, MS, Principal Investigator — Ohio State University
Locations (10):
- United States (10):
  - University of Airzona, Tucson, Arizona
  - Harbor-University of California Los Angeles Medical Center, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of Colordao, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Mecklenburg County Emergency Medical Services, Charlotte, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dell Medical School, University of Texas at Austin, Austin, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bosson N, Hansen M, Gausche-Hill M, Lewis RJ, Wendelberger B, Shah MI, VanBuren JM, Wang HE. Design of a novel clinical trial of prehospital pediatric airway management. Clin Trials. 2022 Feb;19(1):62-70. doi: 10.1177/17407745211059855. Epub 2021 Dec 7. PMID 34875893